CLINICAL TRIAL: NCT06917651
Title: Management of Moderate to Severe Monotraumatic Pain With Sublingual Sufentanil in an Emergency Situation.
Acronym: SubSUF-ER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2024 MOUSTAFA; 2024-519217-64-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
Keywords: pain; sublingual sufentanil; traumatic pain
MeSH Terms: conditions — Agnosia; Pain | interventions — Tablets; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Patient randomized to the "standard of care" arm will receive analgesic treatment according to the department's internal pain management protocol.
  Interventions: Other: Standard of Care (SOC)
- SST 30 mcg (Experimental): Patients randomized to the "SST 30 mcg" arm will receive a 30-microgram sublingual sufentanil tablet.
  Interventions: Drug: sufentanil sublingual 30 mcg tablet

INTERVENTIONS:
Drug: sufentanil sublingual 30 mcg tablet — patient randomized in the "SST 30mcg" arm will receive a 30-microgram sublingual sufentanil tablet
  Arms: SST 30 mcg
Other: Standard of Care (SOC) — patients randomized in the "SOC" arm will receive analgesic treatment according to the department's internal pain management protocol.
  Arms: Standard of Care

SUMMARY:
Pain is a common reason for emergency department (ED) visits. However, studies suggest that emergency physicians may not always provide optimal analgesic treatment due to various factors, such as time constraints, demographic factors like gender and age, and concerns about opioid use. As a result, patients with moderate to severe pain often experience long delays before receiving analgesia and may even be discharged with unresolved pain or suboptimal treatment. Additionally, diagnostic procedures for patients with isolated trauma (e.g., clinical examinations, radiographs) can lead to variations in pain levels, making it difficult to assess the effectiveness of analgesia.

A commonly used treatment for moderate to severe pain is intravenous opioid administration. However, this approach requires longer wait times, complex titration, and significant resources (beds, nurses, equipment), which may be limited during peak hours. While oral opioids require fewer resources, their delayed onset and limited titratability restrict their use for severe pain.

The sublingual sufentanil tablet (30 mcg), delivered via a single-dose applicator, was developed for patients with moderate to severe pain in emergency or outpatient surgical settings. Its unique pharmacokinetic and pharmacodynamic properties could offer advantages in non-invasive acute pain management.

Sublingual sufentanil received market authorization in June 2018 for the treatment of moderate to severe acute pain in adults and is already used in many hospitals. However, further studies are needed to confirm its effectiveness and potential superiority in pain management.

The objective of this study is to evaluate the effectiveness of 30 mcg sublingual sufentanil in patients admitted for moderate to severe pain due to isolated trauma. This will be compared to the standard pain management protocol used in the Clermont-Ferrand emergency department, focusing on pain score variations using a numerical rating scale (0-10)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with a pain rating on the Numerical Rating Scale (NRS) ≥ 4
* Pain of monotraumatic origin in the upper or lower limb
* Glasgow Coma Scale = 15
* SaO2 > 95% in ambient air

Exclusion Criteria:

* Polytrauma
* Analgesic treatment within the 4 hours preceding admission (except paracetamol)
* Woman of childbearing age without effective contraception, declaring pregnancy or at risk of pregnancy, breastfeeding woman, or positive pregnancy test at inclusion
* Patient requiring intravenous access upon admission (e.g., displaced open fracture)
* Contraindication or allergy to any of the molecules in the analgesia protocol
* Refusal to participate
* Known substance abuse or psychiatric disorders
* Known oxygen dependence or COPD
* Not affiliated with social security
* Patient under guardianship, curatorship, deprived of liberty, or under legal protection
* Patient who does not speak or read French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of sublingual sufentanil compared to the standard analgesic protocol used in the department, by measuring pain scores on the Numerical Rating Scale from 0 to 10 at Hour 0 and Hour 0 +60 minutes | Hour 0 ; Hour 0 + 60 minutes
  the efficacy of sublingual sufentanil will be measured by the difference in pain scores measured by the NRS between baseline and 60 minutes after receiving treatment NRS is a 10-point scale where 0 means no pain and 10 means the most pain

SECONDARY OUTCOMES:
Comparison between randomization groups of potential adverse effects. | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  Safety outcomes : The comparison between randomization groups of potential adverse effects: hypotension, bradycardia, respiratory depression, sweating, drowsiness, nausea and/or vomiting, dizziness.
Pain variation assessed at different time points. | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  Pain variation assessed in both groups at different time points of the study. Pain will be evaluated using the NRS, à 10-point scale, where 0 corresponds to no pain and 10 to the most intense pain.
Blood pressure variations | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  Blood pressure variation in patients at different time points, measured using an automatic sphygmomanometer.
Heart rate variations | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  Heart rate variation in patients at different time points, measured using a heart rate monitor.
Oxygen saturation variation | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  Oxygen saturation variation in patients at different time points, measured using a pulse oximeter.
Breath frequency variations | Hour 0 ; Hour 0 + 15 minutes; Hour 0 + 30 minutes; Hour 0 + 45 minutes; Hour 0 + 60 minutes; Hour 0 +120 minutes; Hour 0 + 180 minutes
  variation of breath frequency measured at differents time points
Assessment of patient satisfaction with pain management using a 10-point scale | Hour 0 + 180 minutes
  Assessment of patient satisfaction with pain management using a 10-point scale, where 0 represents "very dissatisfied" and 10 represents "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Farès MOUSTAFA, PR, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France, France

IPD SHARING:
Plan to Share IPD: No